CLINICAL TRIAL: NCT03160274
Title: Genetic Analysis of Pheochromocytomas, Paragangliomas and Associated Conditions
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); The Paradifference Foundation (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSC20060069H; 5R01GM114102 (NIH); R01CA264248-04S2 (NIH)
Record Dates: First submitted 2017-05-05; First posted 2017-05-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Pheochromocytoma; Paraganglioma; Inherited Cancer Syndrome; Associated Conditions; Kidney Neoplasms; Bone Cancer; Thyroid Neoplasms; Other Cancer
Keywords: tumor suppressor gene; oncogene; mutation; susceptibility gene
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Neoplastic Syndromes, Hereditary; Kidney Neoplasms; Bone Neoplasms; Thyroid Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Samples from affected individuals will be obtained as:
  * DNA from peripheral blood lymphocytes,
  * DNA from tumor tissue, or
  * Frozen peripheral blood lymphocytes for nucleic acid purification
  * Frozen tumor tissue for nucleic acid purification
  * Lymphoblastoid cell lines, if available
  * Buccal cells obtained by cheek swab or saliva
  Samples from unaffected relatives will be obtained as:
  * DNA from peripheral blood lymphocytes, or
  * Frozen peripheral blood lymphocytes for nucleic acid purification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Genetic screening — Germline and/or tumor samples will be screened for mutations

SUMMARY:
Pheochromocytomas and paragangliomas are neural crest-derived tumors of the nervous system that are often inherited and genetically heterogeneous. Genetic screening is recommended for patients and their relatives, and can guide clinical decisions. However, a mutation is not found in all cases. The aims of this proposal are to: 1) to map gene(s) involved in pheochromocytoma, and 2) identify genotype-phenotype correlations in patients with pheochromocytoma/paraganglioma of various genetic origins.

DETAILED DESCRIPTION:
Pheochromocytoma and paragangliomas are tumors originated from neuroectoderm cells located in the adrenal or extra-adrenal paraganglia, often leading to increased secretion of hormones known as catecholamines. These tumors represent a potentially curable cause of hypertension and are malignant in about 10-15% of the cases. Approximately 40% of patients with pheochromocytomas and/or paraganglioma have an inherited mutation. In addition, some patients and/or their relatives that are mutation carriers can develop other tumors as part of inherited cancer susceptibility syndromes. Therefore, detection of the susceptibility mutation is important for diagnosis and follow up. However, the susceptibility gene mutation cannot be identified in all cases. Studies that aim to identify novel susceptibility genes for pheochromocytoma are required.

The fist aim of this study is to identify novel pheochromocytoma susceptibility genes. Characterization of such gene(s) can improve our understanding of the pathogenesis pheochromocytoma and paraganglioma and have an impact in diagnosis, therapeutic planning and genetic screening of relatives.

The second aim of this project is to characterize relationships between mutations and clinical features that can provide insights into clinical surveillance and screening of at-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of pheochromocytoma and or paraganglioma
* family member with diagnosis of pheochromocytoma and or paraganglioma
* diagnosis of a pheochromocytoma- and or paraganglioma-associated condition
* family member with diagnosis of a pheochromocytoma- and or paraganglioma-associated condition

Exclusion Criteria:

* unconfirmed diagnosis of pheochromocytoma and/or paraganglioma or associated condition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals must have confirmed personal or family history of pheochromocytoma, paraganglioma or associated conditions. Relatives of patients with pheochromocytoma and/or paraganglioma are also eligible. Consent form will be obtained from all patients. It is expected that a number of participants in the study will be from outside our institution and also outside U.S.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-10-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of germline driver mutation | through study completion- average time approximately 6 months
  Genetic screen detects a mutation that is likely responsible for tumor development
Identification of somatic driver mutation | through study completion- average time approximately 6 months
  Genetic screen detects a mutation that is likely responsible for tumor development

SECONDARY OUTCOMES:
Identification of additional, potentially pathogenic genetic variants | through study completion- average time approximately 6 months
  Genetic screen detects other mutations with potential pathogenic effects
Identification of clinical features other than pheochromocytoma and/or paraganglioma that segregate with disease | through study completion- average time approximately 6 months
  Clinical data reveals other features that might associate with the main disease phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Dahia, MD, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be available in the form of publications and pertinent data will be deposited in public depositories

REFERENCES:
- [Background] Dahia PL. Pheochromocytoma and paraganglioma pathogenesis: learning from genetic heterogeneity. Nat Rev Cancer. 2014 Feb;14(2):108-19. doi: 10.1038/nrc3648. Epub 2014 Jan 20. PMID 24442145